CLINICAL TRIAL: NCT04784624
Title: Virtual Lifestyle Programming to Limit Collateral Health Damage From COVID 19 Pandemic: an Evaluation
Brief Title: Virtual Lifestyle Program Evaluation During Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Seven Oaks Hospital Chronic Disease Innovation Centre (Network)
Responsible Party: Principal Investigator, Claudio Rigatto, Associate professor, University of Manitoba
Other Study IDs: HS24424(H2020:495)
Record Dates: First submitted 2021-02-08; First posted 2021-03-05 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Cardiometabolic Syndrome; Weight Loss
Keywords: virtual platform; evaluation; diet; physical activity; behavior change; sleep; stress
MeSH Terms: conditions — Metabolic Syndrome; Weight Loss; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle program — The cardiometabolic and weight loss program is based on The Wellness Institute clinically validated lifestyle medicine program and will be delivered virtually using a digital platform and artificial intelligence that is supported by a health coach. The program focuses on building individual's self-efficacy, motivation and importance to make and sustain healthy choices. The 16-week program begins with a health risk assessment and a personalized wellness plan. The plan includes a personalized exercise plan and nutrition strategy. Each user will regularly check-in with their personal health coach whose role is to provide expert advice and also empower, support and help make the user accountable as they build a healthy lifestyle. Coaching includes identifying obstacles to changing behaviors and how to develop new behaviors that will become the norm.

SUMMARY:
This is a pilot study evaluating an online cardiometabolic and weight loss program which is offered by The Wellness Institute. The program is 16 weeks and is developed by a multidisciplinary team and delivered by a degreed health professional (health coach) to assist participants in achieving their personal wellness goals. This study will also investigate the impact of Coronavirus Disease (COVID-19) on participants lifestyles and access to lifestyle programs and supports.

DETAILED DESCRIPTION:
The Wellness Institute is offering a new cardiometabolic and weight loss program. It is a digital behavior change program designed to help clients achieve healthy weight reduction, thereby improving cardiometabolic risk. The target population is overweight or obese individuals at risk for or living with health conditions such as pre-diabetes, diabetes, hypertension and high cholesterol. The purpose of this study is to evaluate the program following a mixed methods quasi-experimental approach using focus groups, questionnaires, and data collected over the 16 week duration of the program. Participants will be asked to fill in a set of questionnaires to measure physical activity, diet, sleep and stress at the start and end of the program. Other outcomes include changes in body weight, body mass index (BMI), blood pressure, clinical chemistry, and medication intake over the 16 week program. At the end of the program, adherence will be measured though attendance and platform usage and acceptability will be measured by an exit questionnaire and virtual focus groups. This study will investigate the impact of COVID-19 on participants lifestyles and access to lifestyle programs and support. The impact of COVID-19 will be assessed through a Covid-19 questionnaire and virtual focus groups.

ELIGIBILITY:
Program inclusion criteria:

• Male or female, aged 18 years or above, have one or more of the following conditions: pre-diabetes, diabetes, high blood pressure, high triglycerides, low HDL, abdominal obesity, and BMI >25 kg/m2.

Program exclusion criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the program.
* Recent heart attack, stroke, heart surgery, and congestive heart failure.
* Participants who have unmanaged diabetes, chest pain or difficulty breathing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from individuals enrolled in the online program and willing and able to give informed consent for participation in the evaluation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Impact of COVID-19 survey | Start of the program - first week of enrollment
  A COVID-19 wellbeing survey will be used to understand the impact of COVID-19 pandemic on lifestyle behaviours and programs and services have changed in response to COVID-19
Program adherence | 16 weeks
  Participants will be qualified as adhering to the program if they attend a minimum of 3 out of 4 health coaching sessions and have at least 1 activity during weeks 12-18.

SECONDARY OUTCOMES:
Physical activity level - International Physical Activity Questionnaire-Long (IPAQ-L) | 16 weeks
  International Physical Activity Questionnaire-Long (IPAQ-L) will be used to evaluate participant's physical activity level for the last 7 days at the start and end of program. It comprises a set of 4 questionnaires and 5 activity domains asked independently. This questionnaire assesses the types of intensity of physical activity and the amount of sitting time that people do as part of their daily lives. These are used to estimate total physical activity in MET-min/week and time spent sitting.
Physical activity level - International Physical Activity Questionnaire-Short (IPAQ-S) | 16 weeks
  International Physical Activity Questionnaire-Short (IPAQ-S) will be used to evaluate participant's physical activity level for the last 7 days at the start and end of program. It comprises a set of 4 questionnaires and 4 generic items. This questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives. These are used to estimate total physical activity in MET-min/week and time spent sitting.
Dietary intake | 16 weeks
  Automated Self-Administered Recall System (ASA24) 3-day food recall will be used as tool to recall 3 days of dietary intake at the start and end of program.
Dietary behavior | 16 weeks
  Three factor questionnaire will evaluate changes in participant's dietary habits at the start and end of program. It measures 3 dimensions of human eating behavior: cognitive restraint of eating, disinhibition and hunger.
Dietary habits | 16 weeks
  Mindful eating questionnaire will evaluate changes in participant's dietary behaviors at the start and end of program. It evaluates emotional and behavioral eating habits in designated populations. A higher score may indicate better outcome in long term body weight maintenance.
Sleep | 16 weeks
  Pittsburgh sleep quality index (PSQI) questionnaire will be used to evaluate changes in sleep at the start and end of program. The PSQI is used to measure the quality and patterns of sleep in adults. It includes seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. A score of 5 or less is indicated as good sleep quality where a score of 6 or more is indicated as poor sleep quality.
Stress | 16 weeks
  Perceived stress questionnaire (PSQ) will be used to evaluate changes in stress at the start and end of program. The PSQ is developed as an instrument for assessing the stressful life events and circumstances that tend to trigger or exacerbate disease symptoms.
High-density lipoprotein Cholesterol (HDL-C) | 16 weeks
  HDL-C will be measured at the start and end of program.
Total cholesterol | 16 weeks
  Total cholesterol will be measured at the start and end of program.
Low-density lipoprotein cholesterol (LDL-C) | 16 weeks
  LDL-C will be measured at the start and end of program.
Triglycerides | 16 weeks
  Triglycerides will be measured at the start and end of program.
Total cholesterol/HDL ratio | 16 weeks
  Total cholesterol/HDL ratio will be measured at the start and end of program.
Fasting blood glucose | 16 weeks
  Fasting blood glucose will be measured at the start and end of program.
Insulin | 16 weeks
  Insulin will be measured at the start and end of program.
Hemoglobin A1C | 16 weeks
  Hemoglobin A1C will be measured at the start and end of program.
Body weight | 16 weeks
  Body weight will be measured at the start and end of program.
BMI | 16 weeks
  BMI will be measured at the start and end of program.
Systolic blood pressure | 16 weeks
  Systolic blood pressure will be measured in triplicate the start and end of program.
Diastolic blood pressure | 16 weeks
  Diastolic blood pressure will be measured in triplicate the start and end of program.
Medication intake | 16 weeks
  Participant's medication intake will be tracked and assessed the start and end of program.
Cardiovascular assessment | 16 weeks
  Framingham score will be used to assess participant's 10-year risk of cardiovascular disease the start and end of program.
Impact of COVID-19-focus groups | First 3 months of program initiation
  Focus groups will be conducted with a subset of participants to understand the impact of the COVID-19 pandemic on lifestyle behaviors and on how individuals' needs and perspectives on lifestyle programs and services have changed in response to COVID-19
Program acceptability - exit survey | Program completion at 16 weeks
  A study exit survey will be used to evaluate the program acceptability.
Program acceptability - focus groups | Within 3 months of completing the program
  Focus groups will be conducted with a subset of participants after completion of the program to obtain feedback.
Evaluate participant's program engagement and learning | At the end of the study
  Participant's involvement will be assessed by measuring participant learning and engagement. Participant learning will be measured by the proportion of the workbook steps completed and review of health library educational materials. Engagement in the program will be estimated by the average activity participants engaged in per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Chronic Disease Innovation Centre, Seven Oaks Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Dandeneau D, Leon S, Cameranesi M, Alexiuk M, Protudjer J, Bohm C, DiNella M, Solmundson C, Talson M, Wang H, Whitlock R, Rigatto C, Mollard RC. Evaluation of an online cardiometabolic and weight loss program: a mixed methods study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-11. doi: 10.1139/apnm-2024-0190. PMID 39854690